CLINICAL TRIAL: NCT01676207
Title: Prevalence of Extracardiac Coronary Collateral Supply Via the Internal Mammary Arteries
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 007/12
Record Dates: First submitted 2012-08-28; First posted 2012-08-30 (Estimated); Last update posted 2014-01-16 (Estimated); Status verified 2014-01

CONDITIONS: Coronary Artery Disease; Collateral Circulation; Ischemia
Keywords: coronary collateral circulation; extracardiac coronary collaterals; coronary artery disease; coronary circulation; internal mammary artery
MeSH Terms: conditions — Coronary Artery Disease; Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: CAD
  Interventions: Procedure: Coronary Angiography with collateral flow measurements
- 2: no CAD
  Interventions: Procedure: Coronary Angiography with collateral flow measurements

INTERVENTIONS:
Procedure: Coronary Angiography with collateral flow measurements — * Diagnostic coronary angiography and LV angiography
  * Administration of 5'000 units of heparin i.v. and 2 puffs of oral isosorbide-dinitrate
  * Right and left IMA CFI during a 1-minute ostial vessel occlusion
  * Selection of the coronary artery for CFI according to stenotic lesion chosen for PCI or according to ease of access by the pressure sensor wire. Placement of a non-sensor wire in the left IMA. Two coronary CFI measurements (1-minute occlusion): the first with, the second without distal IMA balloon occlusion. Placement of a non-sensor wire in the right IMA. Two coronary CFI measurements: the first with, the second without distal IMA balloon occlusion.
  * IMA angiography (left and right) during distal IMA and coronary occlusion.
  Groups: 1
Procedure: Coronary Angiography with collateral flow measurements — * Diagnostic coronary angiography and LV angiography
  * Administration of 5'000 units of heparin i.v. and 2 puffs of oral isosorbide-dinitrate
  * Right and left IMA CFI during a 1-minute ostial vessel occlusion
  * Selection of the coronary artery for CFI according to stenotic lesion chosen for PCI or according to ease of access by the pressure sensor wire. Placement of a non-sensor wire in the left IMA. Two coronary CFI measurements (1-minute occlusion): the first with, the second without distal IMA balloon occlusion. Placement of a non-sensor wire in the right IMA. Two coronary CFI measurements: the first with, the second without distal IMA balloon occlusion.
  * IMA angiography (left and right) during distal IMA and coronary occlusion.
  Groups: 2

SUMMARY:
In contrast to the extensively studied coronary collateral circulation within the heart, clinical attention has been paid only anecdotally to extracardiac-to-coronary anastomoses. Usually this has been in the form of case reports giving account of angiographically visible anastomoses between the coronary circulation and the internal mammary artery (IMA), typically in the presence of a chronic occlusion of a coronary artery. In the anatomical literature,the most common types of extracardiac anastomoses include bronchial-to-coronary-artery and IMA-to-coronary-artery connections. Anastomoses between the IMA and the coronary circulation have been documented to occur in 12% of post-mortem patients with CAD.

Importantly, hitherto existing observations typically have relied on visual methods insensitive for the adequate detection especially of structurally present but poorly functional anastomoses. On a diagnostic coronary angiogram, collaterals are visible only if the recipient vessel is subtotally stenotic or fully occluded, or can be rendered visible during coronary spasm or by temporary balloon occlusion of the recipient artery and simultaneous injection of contrast medium into the other arteries, respectively. Similarly, the macroscopic pathologic postmortem examination is likely to underestimate the true number of extracardiac coronary collaterals.

The purpose of this study is to determine the in vivo prevalence and functional distribution of IMA-to-coronary collateral supply via both the right and the left coronary artery.

DETAILED DESCRIPTION:
Background

Surgical bypass creates an artificial anastomosis between a diseased coronary artery and an extracardiac vessel. Often one of the internal mammary arteries (IMA) is used for this procedure. These connections have been very rarely described to occur naturally, representing extracardiac coronary collaterals.

In contrast to the extensively studied coronary collateral circulation within the heart, clinical attention has been paid only anecdotally to extracardiac-to-coronary anastomoses. Usually this has been in the form of case reports giving account of angiographically visible anastomoses between the coronary circulation and the internal mammary artery (IMA), typically in the presence of a chronic occlusion of a coronary artery. In the anatomical literature,the most common types of extracardiac anastomoses include bronchial-to-coronary-artery and IMA-to-coronary-artery connections. Anastomoses between the IMA and the coronary circulation have been documented to occur in 12% of post-mortem patients with CAD.

Importantly, hitherto existing observations typically have relied on visual methods insensitive for the adequate detection especially of structurally present but poorly functional anastomoses. On a diagnostic coronary angiogram, collaterals are visible only if the recipient vessel is subtotally stenotic or fully occluded, or can be rendered visible during coronary spasm or by temporary balloon occlusion of the recipient artery and simultaneous injection of contrast medium into the other arteries, respectively. Similarly, the macroscopic pathologic postmortem examination is likely to underestimate the true number of extracardiac coronary collaterals.

When present, pre-existing connections between the IMA and the coronary circulation could be promoted to serve as natural bypasses to diseased coronary arteries. Promotion of extracardiac blood flow to the coronary circulation has very rarely already been attempted in the past. In a minimally invasive intervention, bilateral surgical ligation of both IMA was performed in a few patients, resulting in clinical improvement and disappearance of angina. However, with the advent of coronary surgery, efforts aimed at promotion of naturally existing bypasses have been abandoned for the placing of artificially created extracardiac anastomoses to the coronary circulation.

Yet with the limitations of these established revascularization interventions becoming clear, the need to search for alternative treatment options gets evident. Therapeutic arteriogenesis with promotion of naturally existing bypasses between the coronary circulation and the internal mammary arteries presents a future possibility.

Objective

The purpose of this study is to determine the in vivo prevalence and functional distribution of IMA-to-coronary collateral supply via both the right and the left coronary artery.

Methods

Comparative observational study with CFI measurements in the IMAs (proximal IMA occlusion) and in the coronary circulation (distal IMA occlusion), and IMA angiography during distal IMA occlusion.

Study Protocol

* Diagnostic coronary angiography and LV angiography
* Administration of 5'000 units of heparin i.v. and 2 puffs of oral isosorbide-dinitrate
* Right and left IMA CFI during a 1-minute ostial vessel occlusion
* Selection of the coronary artery for CFI according to stenotic lesion chosen for PCI or according to ease of access by the pressure sensor wire. Placement of a non-sensor wire in the left IMA. Two coronary CFI measurements (1-minute occlusion): the first with, the second without distal IMA balloon occlusion. Placement of a non-sensor wire in the right IMA. Two coronary CFI measurements: the first with, the second without distal IMA balloon occlusion.
* IMA angiography (left and right) during distal IMA and coronary occlusion.

ELIGIBILITY:
Inclusion Criteria:

* age > 17 years
* electively referred for coronary angiography
* written informed consent to participate in the study

Exclusion Criteria

* Acute coronary syndrome
* Prior coronary artery bypass grafting
* Severe cardiac valve disease
* Congestive heart failure NYHA III-IV
* Severe pulmonary artery hypertension
* Severe hepatic or renal failure (creatinine clearance < 15ml/min)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients electively referred for coronary angiography
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2012-07; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Coronary Collateral Flow Index (CFI) | during coronary artery balloon occlusion

SECONDARY OUTCOMES:
Intra-coronary occlusive ECG ST segment shift (mV) | at 1 minute of coronary artery balloon occlusion
angiographic visibility of coronary collateral supply via the internal mammary artery during their distal balloon occlusion | at 1 minute of coronary artery balloon occlusion

CONTACTS AND LOCATIONS:
Overall Officials: Christian Seiler, MD Prof, Principal Investigator — Department of Cardiology, Bern University Hospital
Locations (1):
- Department of Cardiology, Bern University Hospital, Bern, Switzerland

REFERENCES:
- [Derived] Stoller M, de Marchi SF, Seiler C. Function of natural internal mammary-to-coronary artery bypasses and its effect on myocardial ischemia. Circulation. 2014 Jun 24;129(25):2645-52. doi: 10.1161/CIRCULATIONAHA.114.008898. Epub 2014 Apr 17. PMID 24744276